CLINICAL TRIAL: NCT01478139
Title: Ligation of Intersphincteric Fistula Tract (LIFT) Versus LIFT-plug Procedure for Anal Fistula Repair: a Multicenter, Randomized, Open-label, Parallel Controlled Trial
Brief Title: Ligation of Intersphincteric Fistula Tract (LIFT) Versus LIFT-plug Procedure for Anal Fistula Repair
Acronym: LIFT-plug
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhen Jun Wang (Other)
Collaborators: Peking University Third Hospital (Other); Tianjin Third Central Hospital (Other); Xi'an Jiaotong University (Other); Shaanxi Provincial People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhen Jun Wang, Clinical Professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIFTplug-110212
Record Dates: First submitted 2011-11-10; First posted 2011-11-23 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Anorectal Fistula; Extracellular Matrix Alteration
Keywords: anorectal fistula; acellular dermal matrix; ligation of intersphincteric fistula tract; ligation of intersphincteric fistula tract and plug; complications of treatment; recurrence
MeSH Terms: conditions — Rectal Fistula; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LIFT (Experimental): Subjects randomized to this arm will receive the ligation of the intersphincteric fistula track (LIFT) procedure
  Interventions: Procedure: LIFT
- LIFT-plug (Experimental): Subjects randomized to this arm will receive the ligation of the intersphincteric fistula track and plug (LIFT-plug) procedure
  Interventions: Procedure: LIFT-plug

INTERVENTIONS:
Procedure: LIFT-plug — Subjects randomized to this arm will receive the ligation of the intersphincteric fistula track and plug (LIFT-plug) procedure
  Arms: LIFT-plug
Procedure: LIFT — Subjects randomized to this arm will receive the ligation of the intersphincteric fistula track (LIFT) procedure
  Arms: LIFT

SUMMARY:
The purpose of this study is to validate the effect of Ligation of Intersphincteric Fistula Tract (LIFT) Versus LIFT-plug procedure for Anal Fistula Repair.

DETAILED DESCRIPTION:
The management of trans-sphincteric anal fistulae of cryptoglandular origin is challenging. The ideal management is to effectively heal the fistula without compromising continence, avoid fistula recurrence, and quick recovery. Ligation of the intersphincteric fistula tract (LIFT) and LIFT reinforced with a bioprosthetic graft (BioLIFT) are two recently reported procedures that showed improved healing results. In the LIFT, Rojanasakul et al proposed to identify the fistula tract in the intersphincteric space and subsequent division and ligation of the tract, and the primary healing rate was 94.4%. The following studies reported slightly lower results, but the recurrence rate was as high as 18% to 28%. Ellis et al subsequently described a modified LIFT procedure (BioLIFT procedure) in which a bioprosthetic was placed in the intersphincteric plane to reinforce the closure of the fistula tract (BioLIFT procedure), and yielded a healing rate of 94% in 31 patients who had a minimum of 1 year of follow-up after their last treatment.

The investigators modified the LIFT procedure by combining LIFT with the technique of anal fistula plug. The bioprosthetic plug was placed into the fistula tract through the opening in the external sphincter to the external opening in the skin after LIFT procedure. The present study was designed to assess the preliminary results of LIFT-Plug technique prospectively.

The purpose of this study is to validate the effect of Ligation of Intersphincteric Fistula Tract (LIFT) Versus LIFT-plug procedure for Anal Fistula Repair.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over eighteen years old or less than 65 years old.
* Able to understand and provide informed consent or have a legally authorized representative capable of providing consent.
* Clinical diagnosis of primary anal fistula categorized as trans-sphincteric fistula tract determined to be of cryptoglandular origin (primary or recurrent).

Exclusion Criteria:

* Presence of horseshoe fistula.
* History of immunosuppression therapy/treatment within previous six months.
* Fistulas with active abscess, infection, or acute inflammation
* History of Choron's Disease
* History of Ulcerative Colitis
* History of HIV or other immune system disease
* History of collagen disease
* History of radiation to the anorectal region
* Allergies to pig tissue or pig products
* Religious or cultural objection to the use of pig tissue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Healing time | 1month, 3 month, 6 month postoperatively

SECONDARY OUTCOMES:
recurrence rate | 1month, 3 month, 6 month postoperatively
postoperative pain | 1month, 3 month, 6 month postoperatively
  The methodology used for the evaluation of postoperative perineal pain severity and relief, is the visual analogue scale (VAS) (1-10). We considered positive a VAS > 4.
fecal incontinence | 1month, 3 month, 6 month postoperatively
complication rates | 1month, 3 month, 6 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jun Wang, M.D., Study Chair — Beijing Chao Yang Hospital
Locations (5):
- China (5):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - Xi'an Jiaotong University College of Medicine, Xi’an, Shanxi
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality